CLINICAL TRIAL: NCT05461534
Title: The Effect of Mindfulness Yoga on Sexual Functioning for Breast Cancer Survivors
Brief Title: Mindfulness Yoga and Sexual Functioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Rui Yan, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CTR20220630
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Sexual Dysfunction
MeSH Terms: conditions — Breast Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: mindfulness yoga (Experimental): an 8-week structured mindfulness yoga program
  Interventions: Behavioral: mindfulness yoga
- Waiting-list control group (No Intervention): provided the 8-week structured mindfulness yoga upon their completion of the study

INTERVENTIONS:
Behavioral: mindfulness yoga — Each mindfulness yoga session will last for 90 minutes and will be conducted in a group format once a week. Each session includes breathing exercise (10 min), mindfulness meditation and body scan (20 min) and yoga practice (60 min).
  Arms: Intervention group: mindfulness yoga

SUMMARY:
Female breast cancer survivors with sexual dysfunction were randomly divided into a mindfulness yoga intervention group and a control group, and the investigators aimed to evaluate the effects of mindfulness yoga on sexual function in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

age 18-65 years; diagnosed with primary breast cancer (stages:T1-T4, N0-N1, M0); individuals who have completed surgery, chemotherapy and radiotherapy (with the exception of immunotherapy and endocrine therapy); without cognitive impairment; diagnosed with sexual dysfunction.

Exclusion Criteria:

without sexual experience; in pregnancy or lactation; individuals with serious cognitive or psychiatric issues (i.e., depression, alcohol dependency, or psychotic disorders); individuals who are illiterate, with hearing disorder or communication difficulties; individuals with other type of tumors or other serious acute or chronic diseases at the time of enrollment; individuals participate in a concurrent medical treatment or nonmedical treatment targeting sexual problems; individuals participate in a concurrent psychotherapy; individuals with experience in mindfulness or yoga.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from sexual activity | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The score change of the Sexual Activity Questionnaire(SAQ).The SAQ consists of 10 items and three subscales. Higher pleasure or discomfort subscale score indicated higher levels of pleasure or discomfort, and habit is a single item (0 'less sexual activity than usual' to 3 'much more sexual activity than usual').
Change from Female sexual function index | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The score change of Female Sexual Function Index (FSFI). FSFI consists of 19 items comprising six domains of sexual function (desire, arousal, lubrication, orgasm, satisfaction, and pain). The total score ranges from 0 to 36. Higher score corresponds to better sexual functioning.
Change from Sexual distress | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The change of The Female Sexual Distress Scale-Revised (FSDS-R).The total score ranges from 0 to 48, and a higher score indicates a higher level of sexual distress.

SECONDARY OUTCOMES:
Change from Body Image | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  Body Image Subscale (BIS) of the European Organization for Research and Treatment of Cancer Quality of Life-Breast Cancer Module (EORTC- QLQ-BR23) will be used. The total score ranges from 4 to 16, and higher score indicates higher level of body image.
Change from Anxiety and Depression | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The Hospital Anxiety and Depression Scale (HADS) will be used.Higher HADS-D ( ranges from 0-21) or HADS-A ( ranges from 0-21) score correspond to more serious psychological distress
Change from Menopausal symptoms | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The Endocrine symptom subscale (ESS) of the Endocrine Subscale for The Functional Assessment of Cancer Therapy-Breast (FACT-B ES) will be used. The total score ranges from 0 to 72. Higher score indicates fewer menopausal symptoms
Change from Fatigue | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The Brief Fatigue Inventory (BFI) will be used. The total score ranges from 0 to 90. Higher scores on the BFI indicates greater self-reported levels of fatigue.
Change from Sleep quality | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The Pittsburgh Sleep Quality Index (PSQI) will be used. The total score ranges from 0 to 21. Higher scores indicate poorer sleep quality.
Change from Quality of life (QOL) | 4 weeks (T1), 8 weeks (T2);three months (T3) and six months (T4) after completion of the 8 weeks intervention
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30 (EORTC QLQ-C30) simplified Chinese V3.0 version will be used. The total score ranges from 0 to 100. Higher scores of symptom and financial scales indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

REFERENCES:
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669